CLINICAL TRIAL: NCT02008734
Title: Randomized Short-term Pre-surgical Study to Assess the Effects of PD 0332991 in Early Breast Cancer Patients
Brief Title: Randomized Phase II Study to Assess PD 0332991 in Breast Cancer
Acronym: POP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-002967-24; 2013/2016 (Other: CSET number)
Record Dates: First submitted 2013-12-02; First posted 2013-12-11 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Untreated Operable Early Breast Cancer
MeSH Terms: interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention)
- PD0332991 (Experimental): Patients will be randomized 3:1 to be treated with PD0332991 125mg/day orally for a total duration of 14 days (or 100 mg/day for a total duration of 21 days depending on results of interim analysis) with last treatment taken the day previous to the surgical procedure.
  Interventions: Drug: PD0332991

INTERVENTIONS:
Drug: PD0332991
  Arms: PD0332991

SUMMARY:
This is a Phase II study trying to identify whether short term treatment with PD0332991 yields anti-proliferative response -defined by a low level of Ki67 expression (IHC) at surgery- or induces senescence as determined by SABG expression (IHC) in tumors from patients with early breast cancer non-candidates for neoadjuvant hormonotherapy or chemotherapy, as compared to no treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Female patients aged 18 years or older.
3. Histologically or cytologically confirmed untreated invasive carcinoma of the breast irrespective of HER2 and ER status
4. No personal history of breast cancer within the last 5 years
5. Candidates for initial breast surgery, with a minimum size of 15 mm measured by breast US. Bilateral and multifocal tumors are allowed, assuming tumor evaluations and pre- and post-treatment biopsies are performed in the same target lesion.

7. High proliferative tumor as defined by either Grade 3 or Ki67 ≥20% 8. No evidence of metastatic disease. 9. Eastern Cooperative Oncology Group (ECOG) performance status 0/1. 10. Left ventricular ejection fraction (LVEF) of at least 50% 11. Negative pregnancy test in women of childbearing potential within 14 days prior to treatment initiation (premenopausal or less than 12 months of amenorrhea post-menopause, and who have not undergone surgical sterilization).

12. For women of childbearing potential who are sexually active, agreement to use a highly effective, non-hormonal form of contraception or two effective forms of non-hormonal contraception during and for at least 6 months post-treatment.

13. Patients must be affiliated to a social security system

Exclusion Criteria:

1. Patients non-candidate for upfront breast surgery or candidate for neoadjuvant chemotherapy or hormonotherapy.
2. Patients with previously treated breast cancer during the last 5 years or receiving another concomitant anticancer treatment like chemotherapy, immunotherapy, endocrine

4. Known hypersensibility to PD0332991 or any of its components. 5. Difficulty to swallow oral medication 6. Serious uncontrolled concomitant disease that would put the patient at high risk for treatment-related complications.

7. Patient whose general clinical condition does not consider postponing surgery 8. Inadequate organ function, evidenced by the following laboratory results:

* Absolute neutrophil count <1,500 cells/mm3
* Platelet count <100,000 cells/mm3
* Hemoglobin <9 g/dL
* Total bilirubin greater than 1,5 times the upper limit of normal (ULN) (unless the patient has documented Gilbert's syndrome)
* Aspartate aminotransferase (AST [SGOT]) or alanine aminotransferase (ALT [SGPT]) >2.5 x ULN
* Serum creatinine >2.0 mg/dL and/or 177 μmol/L clearance creatinine <50mL/min (calculated by Cockcroft-Gault method)
* International normalized ratio (INR) and activated partial thromboplastin time (aPTT) or partial thromboplastin time (PTT) >1.5 x ULN (unless on therapeutic coagulation) 9. Uncontrolled hypertension (systolic >150 mmHg and/or diastolic > 100 mmHg) or clinically significant (i.e. active) cardiovascular disease: cerebrovascular accident/stroke or myocardial infarction within 6 months prior to first study medication; unstable angina; CHF of New York Heart Association (NYHA) Grade II or higher; or serious cardiac arrhythmia requiring medication.

  10. Patients with a history of long-QT syndrome or documented family history of long-QT syndrome.

  11. QTc >470 12. serum potassium level < LLN 13. Uncontrolled intercurrent illness including but not limited to, known active infection with human immunodeficiency virus (HIV), hepatitis B or C virus or psychiatric illness/social situations that would limit compliance with study requirements.

  14. Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

  15. Pregnant or breastfeeding patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Anti proliferative response | Assessed at Day 15 after randomization
  percentage of patients who at Day 15 have a natural logarithm of percentage positive IHC staining Ki67 of <1 for each study drug (Ki67 "absolute" antiproliferative responders).

SECONDARY OUTCOMES:
Dose Limiting Toxicity | Assessed at Day 8 and 15 after randomization
  Using NCI CTCAE 4.0
Ki67 | Assessed at Day15 after randomization
  Relative change from baseline to surgery in Ki67 IHC expression ("relative" antripoliferative responders)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Arnedos, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy, Villejuif, Val de Marne, France

REFERENCES:
- [Derived] Turner NC, Liu Y, Zhu Z, Loi S, Colleoni M, Loibl S, DeMichele A, Harbeck N, Andre F, Bayar MA, Michiels S, Zhang Z, Giorgetti C, Arnedos M, Huang Bartlett C, Cristofanilli M. Cyclin E1 Expression and Palbociclib Efficacy in Previously Treated Hormone Receptor-Positive Metastatic Breast Cancer. J Clin Oncol. 2019 May 10;37(14):1169-1178. doi: 10.1200/JCO.18.00925. Epub 2019 Feb 26. PMID 30807234
- [Derived] Arnedos M, Bayar MA, Cheaib B, Scott V, Bouakka I, Valent A, Adam J, Leroux-Kozal V, Marty V, Rapinat A, Mazouni C, Sarfati B, Bieche I, Balleyguier C, Gentien D, Delaloge S, Lacroix-Triki M, Michiels S, Andre F. Modulation of Rb phosphorylation and antiproliferative response to palbociclib: the preoperative-palbociclib (POP) randomized clinical trial. Ann Oncol. 2018 Aug 1;29(8):1755-1762. doi: 10.1093/annonc/mdy202. PMID 29893769
- See also: Related Info — http://www.gustaveroussy.fr/fr/essai/cancers-du-sein-cancer-9